CLINICAL TRIAL: NCT02990195
Title: Restoring the Beneficial Effects of Enterohepatic Bile Salt Signalling by Chyme Reinfusion in Patients With a Double Enterostomy
Acronym: RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC16_8914_RESCUE
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Double Enterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Double enterostomy (Other)
  Interventions: Other: Chyme reinfusion

INTERVENTIONS:
Other: Chyme reinfusion

SUMMARY:
Multicentre prospective human experimental study to determine the effect of chyme reinfusion in patients with a double enterostomy on plasma levels of Fibroblast Growth Factor (FGF19)

DETAILED DESCRIPTION:
Patients supported by chyme reinfusion will be followed for 3 days pre chyme reinfusion and for 7 weeks during chyme reinfusion. Three days prior chyme reinfusion, baseline characteristics will be determined, an ileal biopsy, blood, chyme and urine will be collected. Furthermore, blood, chyme, faeces and urine will be collected at the first day of chime reinfusion. These materials will be collected again at week 1, 3, 5 and 7 weeks after initiation of chyme reinfusion. A second ileal biopsy will be performed at week 3.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or above 18 years old
* Temporary double enterostomy treated by chyme reinfusion as a routine primary care
* Downstream bowel of at least 25 cm of healthy small bowel, accessible by a stoma, and suitable for chyme reinfusion and ileal biopsy
* In case of enterocutaneous fistula, diagnosis of fistula origin and localization confirmed by additional medical imaging (computerized tomography/fistulography)
* Written informed consent.

Exclusion Criteria:

* Patients with a mental disability
* Pregnancy or lactation
* Hepatocellular carcinoma
* Blood coagulation disorders
* Shock of any cause
* Patients subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Effect of chyme reinfusion in patients with a double enterostomy on plasma levels of FGF19 | Week 7

SECONDARY OUTCOMES:
Effect of chyme reinfusion in patients with a double enterostomy on plasma bile salt levels | Week 7
  Measurement of bile salt
Assessment of 7-alpha-hydroxy-4-cholesten-3-one (C4) plasma levels | Week 7
Assessment of bile salt composition in plasma | Week 7
Assessment of microbiotic profiling | Week 7
Assessment of citrulline plasma levels | Week 7
Assessment of intestinal-fatty acid binding protein (I-FABP) plasma levels | Week 7
Assessment of smooth muscle specific (SM) 22 plasma levels | Week 7
Effect of chyme reinfusion in patients with a double enterostomy on liver function | Week 7
Assessment of lipopolysaccharide binding protein (LBP) plasma levels | Week 7
Assessment of plasma levels of inflammatory cytokines interleukin-6 (IL-6) | Week 7
Assessment of plasma levels of tumor necrosis factor-alpha (TNF-alpha) | Week 7

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - CHU de Rennes, Rennes
  - Clinique Saint Yves, Rennes
- Maastricht University, Research Laboratories at the Department of General Surgery, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koelfat KVK, Picot D, Chang X, Desille-Dugast M, van Eijk HM, van Kuijk SMJ, Lenicek M, Layec S, Carsin M, Dussaulx L, Seynhaeve E, Trivin F, Lacaze L, Thibault R, Schaap FG, Olde Damink SWM. Chyme Reinfusion Restores the Regulatory Bile Salt-FGF19 Axis in Patients With Intestinal Failure. Hepatology. 2021 Nov;74(5):2670-2683. doi: 10.1002/hep.32017. Epub 2021 Aug 26. PMID 34133768